CLINICAL TRIAL: NCT02943538
Title: Clinical Impact of Telemedicine in Crohn's Disease and Ulcerative Colitis: Study Teccu
Brief Title: Telemedicine Crohn's Disease and Ulcerative Colitis (TECCU)
Acronym: TECCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Study Teccu
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Crohn's Disease; Colitis, Ulcerative
Keywords: Crohn's Disease; Colitis, Ulcerative; Telemedicine
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telemedicine group (Experimental): In this group, monitoring and control is performed through telematics platform integrated management of chronic NOMHAD, configurated to respond the patients specific needs.
  Interventions: Device: Telemedicine
- Telephone support group (Experimental): A telephone control of their state and evolution will be made through the nursing staff of the unit.
  Interventions: Device: Telephone
- Control group (Active Comparator): Conventional care provided in the unit to patients with IBD -high moderate complexity.
  Interventions: Other: Conventional care

INTERVENTIONS:
Device: Telemedicine — Monitoring and control is performed through telematics platform integrated management of chronic NOMHAD, configurated to respond the patients specific needs.
  Arms: Telemedicine group
Device: Telephone — A telephone control of their state and evolution will be made through the nursing staff of the unit.
  Arms: Telephone support group
Other: Conventional care — Conventional care provided in the unit to patients with IBD -high moderate complexity.
  Arms: Control group

SUMMARY:
Pragmatic clinical trial, randomized, controlled parallel, 3 group (group technology platform, call group and control group), developed in the monograph Reference Unit of Inflammatory Bowel Disease Valencia (single-center).

DETAILED DESCRIPTION:
Hypothesis: The interventions follow-up of patients with Crohn's Disease or Ulcerative Colitis active moderate-high complexity based on the incorporation of information technologies and communication, to improve monitoring of the presence of inflammatory activity, adherence to treatment and drug toxicity, increase the proportion of inactive patients (clinical remission) at 6 months follow-up and thus improve clinical outcomes and health outcomes (HRQOL, satisfaction) and reduces the consumption of health resources.

Goals:

* Primary: To assess the effectiveness of intervention Teccu to achieve clinical remission of IBD patients with moderate-high compared to usual care to these patients (G_control) and assisted call with nurses (G_AT) complexity.
* Secondary: - To evaluate the effectiveness of interventions to improve HRQOL and satisfaction with treatment in patients GTECCU intervention group compared to G_control and G_AT in the 6 months follow up. - To assess the safety of the intervention Teccu judging by adverse events that require a doctor's visit or unscheduled nursing. - Describe the use of health resources (surgeries, hospitalizations, emergency room visits and outpatient visits) by patients of G-Teccu, G_control and G_AT in the 6 months follow up. - Evaluate the effectiveness of intervention in the reduction of a combined endpoint of hospital emergency room visits and unscheduled patients in the intervention group compared to G-Teccu G_control and G_AT within 6 months of follow-up consultations.

Description:

The proposed intervention is based on the extent of chronic GeCronic program that is currently being developed at the Hospital La Fe de Valencia for comprehensive management of chronic conditions of high complexity using the technology platform NOMHAD. NOMHADchronic is a system designed to allow management services to deploy chronically ill supported by technology. The product consists of different modules that seek to cover all aspects of that management: clinical information on the status of patients according to their respective conditions, support for the coordination of the actors during the care process, logistics management and human resources, integration with accessories and monitoring devices. Of all the modules of the platform, NOMHADcore out as the module which houses all the functionality on clinical and care management of patients. There follows a detailed description of the module, its structure and operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Inflammatory Bowel Disease at least 6 months duration, diagnosed according to the classical criteria of Lennard-Jones
* Patients with Crohn's Disease or Ulcerative Colitis with moderate or severe activity (as Harvey-Bradshaw index and May, respectively) attending IBD unit during the period of inclusion.
* Patients who initiate medical treatment with immunosuppressive drugs or biological agents, or are undergoing surgical treatment (surgery is considered as a treatment for EC).
* Patient consents to participate in the study and sign and date personally indicating that it has been informed of all pertinent aspects of the study.
* Patient not incur the exclusion criteria

Exclusion Criteria:

* Patients with cognitive or sensory impairments or with insufficient command of the two official languages of Valencia, in the opinion of the health professional conduct recruitment, hinder the understanding of the issues raised in the surveys, scales or instruments used in the study always who do not have a legal representative
* Patients who are unable to handle a mobile phone to participate in the study. - Patients who do not have a phone line because, if they are assigned to G_TECCU or G_AT groups could not be implemented appropriate interventions.
* They are participating at the time of recruitment in any other clinical trial or experimental study. Exclusion criteria will not be participating in observational studies
* Terminals and / or palliative care according to the criteria of the SECPAL (Spanish Society of Palliative Care) Patients
* Patients institutionalized
* They are members of the research team, the staff of the research center or health centers involved in the study, or any other person directly involved in the study.
* Relatives in the first degree of consanguinity or affinity of members of the research team, the staff of the research center or health centers involved in the study, or any other person directly involved in the study
* Patients presenting as primary diagnosis mental illness
* Patients with active cancer diagnosis
* Patients in the assessment of professional performing recruitment not considered likely to be included for specific monitoring found in another unit such as hemodialysis, transplant unit, day hospital ...
* Patients who do not agree to participate in the study or not to sign the corresponding informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinical Remission | 6 months
  Clinical remission of patients at 6 months of follow-up using Harvey-Bradshaw index for Crohn's disease.
Clinical Remission | 6 months
  Clinical remission of patients at 6 months of follow-up using May index for ulcerative colitis.

SECONDARY OUTCOMES:
Health-Related Quality of Life | 6 months
  Health-Related Quality of Life measured by the generic Euroqol (EQ-5D) questionaire
Health-Related Quality of Life | 6 months
  Health-Related Quality of Life measured by the specific IBD in its reduced version (SIBDQ: Short Inflammatory Bowel Disease Questionnaire).
Patient Satisfaction | 6 months
  Measured by a satisfaction questionaire designed for the study.
Therapeutic adherence | 6 months
  Measured by the validated Morisky-Green questionaire.
Urgent and scheduled visits and urgent hospital admissions | 6 months
  Urgent and scheduled visits and urgent hospital admissions in the follow-up period will be captured directly systems hospital information (HIS).
Number of surgical interventions related with the pathology | 6 months
Work activity and productivity (Cronh patients) | 6 months
  Worrk activity and productivity measured by a validate questionaire: Vergara M. et al. Value Health 2011;14(6):859-61).
Mortality | 6 months
Directs health costs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marian Aguas, Principal Investigator — Instituto de Investigación Sanitaria La Fe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Hoyo J, Nos P, Bastida G, Faubel R, Munoz D, Garrido-Marin A, Valero-Perez E, Bejar-Serrano S, Aguas M. Telemonitoring of Crohn's Disease and Ulcerative Colitis (TECCU): Cost-Effectiveness Analysis. J Med Internet Res. 2019 Sep 13;21(9):e15505. doi: 10.2196/15505. PMID 31538948
- [Derived] Aguas M, Del Hoyo J, Faubel R, Munoz D, Dominguez D, Bastida G, Navarro B, Barrios A, Valdivieso B, Correcher M, Nos P. A Web-Based Telemanagement System for Patients With Complex Inflammatory Bowel Disease: Protocol for a Randomized Controlled Clinical Trial. JMIR Res Protoc. 2018 Dec 21;7(12):e190. doi: 10.2196/resprot.9639. PMID 30578197
- [Derived] Del Hoyo J, Nos P, Faubel R, Munoz D, Dominguez D, Bastida G, Valdivieso B, Correcher M, Aguas M. A Web-Based Telemanagement System for Improving Disease Activity and Quality of Life in Patients With Complex Inflammatory Bowel Disease: Pilot Randomized Controlled Trial. J Med Internet Res. 2018 Nov 27;20(11):e11602. doi: 10.2196/11602. PMID 30482739